CLINICAL TRIAL: NCT06640062
Title: Evaluation of Ultrasound-Guided Erector Spinae Plane Block Versus Oblique Subcostal Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy: A Comparative Study
Brief Title: Ultrasound-Guided Erector Spinae Plane Block Versus Oblique Subcostal Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Michael Fayez Yousef Metias, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Helwan University, Egypt., Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118-2022
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ultrasound; Erector Spinae Plane Block; Oblique Subcostal Transversus Abdominis Plane Block; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Active Comparator): Patients received ultrasound-guided erector spinae plane block.
  Interventions: Other: Erector spinae plane block
- Oblique subcostal transversus abdominis plane block group (Experimental): Patients received ultrasound-guided oblique subcostal transversus abdominis plane block.
  Interventions: Other: Oblique subcostal transversus abdominis plane block

INTERVENTIONS:
Other: Erector spinae plane block — Patients received ultrasound-guided erector spinae plane block.
  Arms: Erector spinae plane block group
Other: Oblique subcostal transversus abdominis plane block — Patients received ultrasound-guided oblique subcostal transversus abdominis plane block.
  Arms: Oblique subcostal transversus abdominis plane block group

SUMMARY:
The aim of this work was to compare the effect of using oblique subcostal transversus abdominis plane (OSTAP) block and erector spinae plane (ESP) block as a part of multi-modal analgesia technique in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a commonly performed surgery and requires multi-modal analgesia for better control of pain. Untreated post-operative pain has many consequences, including patient dissatisfaction, transition into chronic pain, delayed discharge from the hospital, and increased healthcare costs.

Many inter-fascial plane blocks like oblique subcostal transversus abdominis plane (OSTAP) block and recently, erector spinae plane (ESP) block have been utilized as a part of multi modal analgesia technique in many abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years.
* Both gender.
* American Society of Anesthesiologists (ASA) grade I and II physical status.
* Body mass index (BMI): ≥ 20 kg/m2 and ≤ 35 kg/m2.
* Underwent laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient refusal.
* Known sensitivity or contraindication to drugs used in the study (local anesthetics, opioids).
* History of psychological disorders and/or chronic pain syndrome.
* Contraindication to regional anesthesia, e.g., local sepsis, pre-existing peripheral neuropathies, and coagulopathy.
* Severe respiratory disorders such as (severe obstructive pulmonary disease, forced expiratory volume (FEV1), forced vital capacity (FVC) <50% or severe restrictive pulmonary disease, and adult respiratory distress syndrome).
* Severe cardiac disorders such as (heart failure).
* Advanced liver disease (elevated liver enzymes more than 3 folds of normal range).
* Advanced kidney disease (Decreased creatinine clearance <40 ml/min).
* Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Degree of pain intensity | 24 hours postoperatively
  The degree of pain intensity was assessed using the Visual Analogue Scale (VAS). Each patient was instructed about postoperative pain assessment with the VAS. VAS(0 represents "no pain" while 10 represents "the worst pain imaginable"). It was assessed at 30 minutes, 2, 4, 6, 8, 12, 16, 20, and 24 hours postoperatively.

SECONDARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Time to first rescue analgesia was assessed from the end of surgery to the first dose of morphine administrated
Total amount of morphine consumption | 24 hours postoperatively
  When a patient complains of pain equivalent to the Visual Analogue Scale (VAS) ≥ 3, rescue analgesia is given in the form of morphine (0.05mg/kg) intravenous increments, as needed.
Morphine-related side effects | 24 hours postoperatively
  Morphine-related side effects such as incidence of nausea and vomiting, respiratory depression (respiratory rate < 8 breaths/min), bradycardia (heart rate decreases by > 20% of basal reading), pruritus, and urine retention were recorded.
Local anesthetics-related side effects | 24 hours postoperatively
  Local anesthetics-related side effects such as lightheadedness, circumoral numbness, tongue paresthesia, drowsiness, irritability, muscle twitches, convulsions, bradycardia, hypotension (mean arterial blood pressure decreases by > 20% of basal reading), hypoventilation and cardiac arrest were recorded.
Incidence of adverse effects of the block technique | 24 hours postoperatively
  Signs of adverse effects of the block techniques, such as local site infection, hematoma formation, bowel perforation, or pneumothorax, were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.